CLINICAL TRIAL: NCT07240909
Title: A Multicenter, Randomized, PROBE Trial on Antihypertensive Drug Selection Based on Hemodynamic Phenotypes Defined by Bioelectrical Impedance Analysis
Brief Title: Antihypertensive Drug Selection Based on Hemodynamic Phenotypes
Acronym: HEMOPHENO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R25070
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: hypertension; anti-hypertensive therapy; Hemodynamics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemodynamics-based individualized antihypertensive therapy (Experimental): The antihypertensive strategy is individualized according to the patient's hemodynamic indices:
  High-resistance type: Amlodipine Besylate Tablets 5mg, once daily, orally. High cardiac output type: Metoprolol Sustained-Release Tablets 47.5mg, once daily, orally.
  Hypervolemic type: Indapamide Tablets 2.5mg, once daily, orally.
  Interventions: Drug: hemodynamics-based individualized antihypertensive therapy
- guideline-based conventional therapy (Active Comparator): Developing a monotherapy antihypertensive treatment plan for participants based on the 2024 Chinese hypertension guidelines
  Interventions: Drug: guideline-based conventional treatment

INTERVENTIONS:
Drug: hemodynamics-based individualized antihypertensive therapy — The antihypertensive strategy is individualized according to the patient's hemodynamic indices:
  High-resistance type: Amlodipine Besylate Tablets 5mg, once daily, orally. High cardiac output type: Metoprolol Sustained-Release Tablets 47.5mg, once daily, orally.
  Hypervolemic type: Indapamide Tablets 2.5mg, once daily, orally. Participants will take the therapy for 8 weeks.
  Other Names: individualized therapy
  Arms: hemodynamics-based individualized antihypertensive therapy
Drug: guideline-based conventional treatment — Developing a monotherapy antihypertensive treatment plan for participants based on the 2024 Chinese hypertension guidelines.
  Participants will take this treatment for 8 weeks.
  Other Names: conventional treatment
  Arms: guideline-based conventional therapy

SUMMARY:
The goal of this clinical trial is to explore the clinical efficacy and safety of individualized antihypertensive medication guided by hemodynamic phenotyping. The main questions it aims to answer are:

1. Does hemodynamics-based individualized antihypertensive therapy achieve better blood pressure control compared to guideline-based conventional therapy?
2. Does hemodynamics-based individualized therapy have comparable safety to guideline-based conventional treatment? Researchers will compare hemodynamics-based individualized antihypertensive therapy to guideline-based conventional treatment to see if the former is better than the latter.

Participants will:

1. Take hemodynamics-based individualized antihypertensive therapy or guideline-based conventional treatment every day for 8 weeks
2. Visit the clinic once every 4 weeks for checkups and tests
3. Keep a diary of their symptoms and any treatment

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥30 and <80 years, regardless of gender;
2. Confirmed diagnosis of hypertension meeting the criteria outlined in the 2024 Chinese Hypertension Guidelines: office blood pressure ≥140/90 mmHg and home blood pressure ≥135/85 mmHg;
3. Mild to moderate hypertension, with office blood pressure ranging from 140-179/90-109 mmHg;
4. No prior use of antihypertensive medications;
5. Voluntary participation in the study with written informed consent obtained.

Exclusion Criteria:

1. Diagnosed or highly suspected secondary hypertension;
2. Classified as mixed type according to hemodynamic typing;
3. Allergy to the intended antihypertensive medications;
4. Dysphagia;
5. Pregnant or lactating women;
6. Potential pregnancy plans during the trial period;
7. Uncorrected electrolyte disturbances;
8. Severe organ dysfunction;
9. Comorbid conditions leading to inaccurate blood pressure measurement;
10. Comorbid conditions or states unsuitable for noninvasive hemodynamic measurement via bioelectrical impedance;
11. Comorbid conditions contraindicating or requiring caution with trial medications;
12. Comorbid conditions affecting the absorption, distribution, metabolism, or excretion of trial drugs;
13. Concurrent or planned use of medications contraindicated or requiring caution with trial drugs;
14. Concurrent or planned use of medications interfering with trial outcomes;
15. Clinician's assessment deems the patient unsuitable for the trial's antihypertensive regimen;
16. Current participation in other clinical studies that may interfere with the conduct of this trial.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in office systolic blood pressure reduction | 8 weeks after treatment
  Difference in office systolic blood pressure reduction between two groups.

SECONDARY OUTCOMES:
Reduction difference in office systolic blood pressure | 4 weeks after treatment
  Reduction difference in office systolic blood pressure between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Reduction difference in office diastolic blood pressure | 4 weeks after treatment
  Reduction difference in office diastolic blood pressure between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Reduction difference in office mean blood pressure | 4 weeks after treatment
  Reduction difference in office mean blood pressure between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference in pulse rate changes | 4 weeks after treatment
  Difference in pulse rate changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference in blood pressure target rate | 4 weeks after treatment
  Difference in blood pressure target rate (both systolic and diastolic blood pressure will be measured) between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference of systemic vascular resistance index (SVRI) changes | 4 weeks after treatment
  Difference of systemic vascular resistance index (SVRI) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference of cardiac index (CI) changes | 4 weeks after treatment
  Difference of cardiac index (CI) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference of thoracic fluid content (TFC) changes | 4 weeks after treatment
  Difference of thoracic fluid content (TFC) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Reduction difference in office diastolic blood pressure | 8 weeks after treatment
  Reduction difference in office diastolic blood pressure between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Reduction difference in office mean blood pressure | 8 weeks after treatment
  Reduction difference in office mean blood pressure between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference in pulse rate changes | 8 weeks after treatment
  Difference in pulse rate changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy
Difference in blood pressure target rate | 8 weeks after treatment
  Difference in blood pressure target rate (both systolic and diastolic blood pressure will be measured) between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy
Difference of systemic vascular resistance index (SVRI) changes | 8 weeks after treatment
  Difference of systemic vascular resistance index (SVRI) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference of cardiac index (CI) changes | 8 weeks after treatment
  Difference of cardiac index (CI) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.
Difference of thoracic fluid content (TFC) changes | 8 weeks after treatment
  Difference of thoracic fluid content (TFC) changes between two groups and among subgroups of hemodynamic phenotyping in individualized antihypertensive therapy.

OTHER OUTCOMES:
Adverse events | Eight weeks
  Adverse events between two groups
Serious adverse events | Eight weeks
  Serious adverse events between two groups
Adverse drug reaction | Eight weeks
  Adverse drug reaction between two groups

IPD SHARING:
Plan to Share IPD: Yes
Coded data (without personal identification information) used and analysed during the study will be available to researchers one year after the publication date of the manuscript from the corresponding author on reasonable request, with the approval of the steering committee and Research Center for Clinical Trials of the Third Xiangya Hospital of Central South University, on signing of a data access agreement.
Supporting Information: Study Protocol
Time Frame: One year after the publication date of the manuscript.
Access Criteria: Coded data (without personal identification information) used and analysed during the study will be available to researchers one year after the publication date of the manuscript from the corresponding author on reasonable request, with the approval of the steering committee and Research Center for Clinical Trials of the Third Xiangya Hospital of Central South University, on signing of a data access agreement.
URL: https://gcp.xy3yy.com/lixi/index.html